CLINICAL TRIAL: NCT07109830
Title: Utilizing an Electroencephalography-Based Brain-Computer Interface Game to Evaluate Cognitive Skills in Children With Motor Impairments
Brief Title: Utilizing an EEG-Based BCI Game to Evaluate Cognitive Skills in Children With Motor Impairments
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00153206
Record Dates: First submitted 2025-07-21; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Children With Motor Impairments

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typically developing children
  Interventions: Diagnostic Test: Cognitive assessment; Diagnostic Test: NEPSY-II
- Children with motor impairments
  Interventions: Diagnostic Test: Cognitive assessment

INTERVENTIONS:
Diagnostic Test: Cognitive assessment — Cognitive assessment using BCI-game
Diagnostic Test: NEPSY-II — Standardized cognitive assessment
  Groups: Typically developing children

SUMMARY:
This project aims to validate an EEG-based brain-computer interface (BCI) game as a cognitive assessment tool for children with motor impairments. Traditional cognitive assessments often rely on motor responses, which may underestimate the abilities of children with limited mobility. By using BCI technology, which captures brain activity directly, the study seeks to bypass these limitations and offer a more inclusive, engaging, and accurate assessment method.

The research consists of three papers:

1. Pilot Study: Tests the feasibility of the BCI game, comparing BCI and keyboard controls, and examines alignment with NEPSY-II cognitive subtests.
2. Validation Study: Investigates the convergent validity of the BCI game in typically developing children by correlating game performance with standardized cognitive test scores.
3. Adaptation Study: Compares game performance between neurotypical children and children with motor impairments to evaluate the game's inclusivity and adaptability.

The project utilizes the Emotiv Flex 2 EEG system and focuses on cognitive domains such as attention, working memory, and inhibition. The ultimate goal is to develop a reliable, equitable tool for assessing cognition in children with diverse motor abilities.

ELIGIBILITY:
Inclusion Criteria:

* Children with and without motor impairments.
* Ages 7-16.
* Understand simple commands

Exclusion Criteria:

* Vision impairment

Ages: 7 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Typically developing children and children with motor impairments
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological assessment (NEPSY-II) | "Baseline (Day 1): NEPSY-II will be administered during the single study session at the same visit as the BCI game."
  The NEPSY-II (A Developmental Neuropsychological Assessment, Second Edition) is a standardized cognitive assessment for children aged 3-16 years. It evaluates multiple domains of cognitive functioning, including Attention and Executive Functioning, Memory and Learning, and Visuospatial Processing. Each subtest yields a scaled score ranging from 1 to 19 (mean = 10, SD = 3) and domain-level standard scores (mean = 100, SD = 15). Higher scores indicate better cognitive performance.
BCI game metrics | Baseline (Day 1; during the single study visit)
  The BCI-controlled adventure-style game is designed to assess cognitive domains including attention, working memory, and inhibitory control. Participants navigate a virtual environment by turning left or right using brain-computer interface control based on steady-state visually evoked potentials (SSVEP).
  Coins collected reflect the participant's sustained attention and working memory by requiring consistent focus and memory of task-specific rules (e.g., avoiding certain coin colors).
  Obstacles avoided reflect inhibitory control by requiring participants to suppress automatic responses and adapt to changing task demands.
  Each metric is a count variable (0-maximum possible in the game), where higher values indicate better cognitive performance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Only people working on this project will have access to identifiable information and it will be store in an encrypted file